CLINICAL TRIAL: NCT04823689
Title: Reduction of Anterior Glenohumeral Dislocation in Ventral Decubitus Versus Dorsal Decubitus Under Procedural Sedation : a Prospective Randomized Trial
Brief Title: Reduction of Anterior Glenohumeral Dislocation in Ventral Decubitus Versus Dorsal Decubitus Under Procedural Sedation
Acronym: EPOLUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01 - EPOLUX
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Reduction; Emergencies; Anterior Shoulder Dislocation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dorsal decubitus (Sham Comparator): The dorsal decubitus reduction consists in placing the patient in the dorsal position and achieving reduction by traction maneuvers on the luxated upper limb. This maneuver generally requires procedural sedation. A mild traction of the traumatized limb in the axis is performed, with slight external rotation and progressive abduction. In the absence of reduction at this stage, this gesture is completed by a flexion adduction of the limb. A counterweight is then made by a rolled sheet and passed under the armpit of the patient.
  Interventions: Procedure: reductions
- Ventral decubitus (Experimental): The ventral decubitus reduction consists in placing the patient in the ventral position. The luxated limb is positioned in pendulum and the line of contact with the stretcher must pass through the mid-clavicular line. The humeral head is brought to the scapula.
  Interventions: Procedure: reductions

INTERVENTIONS:
Procedure: reductions — Two reduction techniques are compared: dorsal decubitus and ventral decubitus reduction. The dorsal decubitus reduction consists in placing the patient in the dorsal position and achieving reduction by traction maneuvers on the luxated upper limb. This maneuver generally requires procedural sedation. A mild traction of the traumatized limb in the axis is performed, with slight external rotation and progressive abduction. In the absence of reduction at this stage, this gesture is completed by a flexion adduction of the limb. A counterweight is then made by a rolled sheet and passed under the armpit of the patient.
  The ventral decubitus reduction consists in placing the patient in the ventral position. The luxated limb is positioned in pendulum and the line of contact with the stretcher must pass through the mid-clavicular line. The humeral head is brought to the scapula.

SUMMARY:
The anterior glenohumeral dislocation is frequently encountered in emergency medicine. It represents about 50% of the total dislocation and affects 1 resident for 10 000 in France.

In Nord Franche-Comte Hospital, 1 to 2 patients per day present this diagnosis in the emergency department, which requires reduction by external manoeuvres.

A retrospective study shows the interest of the ventral decubitus compared to dorsal decubitus reduction in the care of patients with anterior glenohumeral dislocation. None prospective study has already demonstrate the interest of the ventral decubitus compared to the dorsal decubitus in the reduction of anterior glenohumeral dislocation.

The main objective is to evaluate the speed of the reduction of the anterior dislocation of the shoulder by the ventral decubitus technique compared to the conventional technique in dorsal decubitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiological confirmed anterior glenohumeral dislocation
* Patient affiliated or entitled to a social security scheme
* Oral informed consent form

Exclusion Criteria:

* Glenohumeral fracture or vasculoneural lesion associated
* Dislocation for more than 12 hours
* Homolateral shoulder surgery antecedent
* Contraindication to other analgesics (morphine, sedation)
* BMI > 40
* Patient < 18 year
* Pregnancy or nursing woment
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
The main objective is to evaluate the speed of the reduction of the anterior dislocation of the shoulder by the ventral decubitus technique compared to the conventional technique in dorsal decubitus. | 1 day
  The primary endpoint is the reduction time in minutes from inclusion of the patient after prior confirmation of the clinical and radiological diagnosis to the observed reduction.

SECONDARY OUTCOMES:
Evaluation of the success rate of the ventral decubitus technique compared to the dorsal decubitus technique | 1 day
  Failure rate of the ventral decubitus technique compared to the dorsal decubitus technique
Evaluation of the consumption of sedative and analgesic treatments | 1 day
  Quantification of doses of analgesics and sedatives used
Evaluation of the time spent in emergency department | 1 day
  Time spent in emergency department
Evaluation of the pain felt before and after the intervention | 1 day
  Pain sensibility before, during et after the reduction techniques : visual analog pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Belfort, France

IPD SHARING:
Plan to Share IPD: No